CLINICAL TRIAL: NCT03582527
Title: The Expression of Programmed Death Ligand-1 (PD-L1) on Advanced Osteosarcoma Tissue and Its Influence on Prognosis
Brief Title: PD-L1 Expression in Advanced Osteosarcoma
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: PKUPH-sarcoma 03
Record Dates: First submitted 2018-06-10; First posted 2018-07-11 (Actual); Last update posted 2018-08-01 (Actual); Status verified 2018-07

CONDITIONS: Progression; Survival
Keywords: osteosarcoma; refractory to chemotherapy; unresectable; PD-L1; VENTANA PD-L1 (SP263)
MeSH Terms: conditions — Disease Progression; Osteosarcoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- observation group: All these patients who have been tested will be observed for further treatment and been recorded for toxicity.
  Interventions: Other: all study participants

INTERVENTIONS:
Other: all study participants — patients will receive anti-PD-1/anti-PD-L1 antibody for further treatment

SUMMARY:
The expression level of PD-L1 on tumor cells is a pivotal point which might have some influence on prognosis, especially for those who might use PD-1 or PD-L1 antibody for treatment. The aim of this study is to detect the expression of PD-1 on advaced osteosarcoma patient who might use these antibodies for treatment. All those specimen should be taken by pathologist and confirmed with high tumor cellularity.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis confirmed histologically and reviewed centrally;
* received surgery in Musculoskeletal Tumor Center of Peking University People's Hospital with appropriate sample for immunohistochemical staining;
* progressing upon prior treatment (completed >4 weeks before trial entry) consisted of standard high-grade osteosarcoma chemotherapy agents including doxorubicin, cisplatin, high-dose methotrexate, and ifosfamide; metastatic relapsed and unresectable progressive disease (PD);
* having measurable lesion according to RECIST 1.1;
* Eastern Cooperative Oncology Group performance status 0-1 with a life expectancy >3 months;
* intend to receive anti-PD-1/anti-PD-L1 antibody for therapy.

Exclusion Criteria:

* fail to be followed up regularly.
* sample disqualification.

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: All those advanced osteosarcoma patients who intend to receive anti-PD-1/anti-PD-L1 therapy.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2018-06-01 (Actual); Primary Completion 2019-12-31 (Estimated); Study Completion 2020-02-15 (Estimated)

PRIMARY OUTCOMES:
PD-L1 expression level | 2 months
  all those specimens will be tested for expression level,Tumors with ≥50% cells showing positive membrane staining were considered to have high expression of PD-L1

SECONDARY OUTCOMES:
progression free survival | 2 years
  from the timing of testing to disease progression/death whichever comes first
overall survival | 5 years
  from the timing of testing to death/last follow-up

CONTACTS AND LOCATIONS:
Locations (1):
- Musculoskeletal Tumor Center of Peking University People's Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No